CLINICAL TRIAL: NCT05164952
Title: Delayed Versus Immediate Use Of Zoledronic Acid For Postmenopausal Patients With ER/PR Positive Early Breast Cancer Who Are Using Adjuvant Letrozole
Brief Title: Delayed Versus Immediate Use Of Zoledronic Acid For Postmenopausal Patients With Early Breast Cancer Who Are Using Adjuvant Letrozole
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MAI MOHAMED HEMMAT ABDELFATAH ABDELGELIL, Assistant Lecturer of Clinical Oncology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zoledronic Acid In Breast Ca
Record Dates: First submitted 2021-10-13; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Use of Zoledronic Acid in Breast Cancer
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Delayed use of zoledronic acid arm (Experimental): delayed-ZOL patients will receive ZOL only if their T-score fall below -2.0, after a nontraumatic clinical fracture, or if an asymptomatic fracture will be detected by spinal X-ray at the 3- monthly assessment.
  Interventions: Drug: Zoledronic Acid 4 MG
- Immediate use of zoledronic acid arm (Experimental): Immediate-ZOL patients will receive ZOL immediately after randomization
  Interventions: Drug: Zoledronic Acid 4 MG

INTERVENTIONS:
Drug: Zoledronic Acid 4 MG — (4 mg via 15-min infusion every 6 months) for 24 months
  Other Names: Zometa

SUMMARY:
The investigators will involve about 25 Patients of postmenopausal women who have ER/PR positive early breast cancer in each arm.

The study is a two-arm comparative, prospective, interventional, and randomized study. All patients who are on oral daily letrozole (2.5 mg), will be randomly assigned to receive either immediate or delayed ZOL (4 mg via 15-min infusion every 6 months) for 24 months. Immediate-ZOL patients will receive ZOL immediately after randomization; delayed-ZOL patients will receive ZOL only if their T-score fall below -2.0, after a nontraumatic clinical fracture, or if an asymptomatic fracture will be detected by spinal X-ray at the 3- monthly assessment. All patients will receive daily supplements containing calcium (500 mg) and vitamin D (400-800 IU). Baseline bone mineral density and every 3 months will be done for the enrolled patients.

DETAILED DESCRIPTION:
The investigators will involve about 25 Patients of postmenopausal women who have ER/PR positive early breast cancer in each arm.

The study is a two-arm comparative, prospective, interventional, and randomized study. All patients who are on oral daily letrozole (2.5 mg), will be randomly assigned to receive either immediate or delayed ZOL (4 mg via 15-min infusion every 6 months) for 24 months. Immediate-ZOL patients will receive ZOL immediately after randomization; delayed-ZOL patients will receive ZOL only if their T-score fall below -2.0, after a nontraumatic clinical fracture, or if an asymptomatic fracture will be detected by spinal X-ray at the 3- monthly assessment. All patients will receive daily supplements containing calcium (500 mg) and vitamin D (400-800 IU). Baseline bone mineral density and every 3 months will be done for the enrolled patients.

-Research outcome measures:

1. Primary (main): The primary endpoint will be the percentage change in lumber spine (L2-L4) BMD at 12 months for immediate- versus delayed-ZOL patients.
2. Secondary (subsidiary): Secondary end points will include percentage change in total hip BMD at each assessment, fracture incidence, time to disease recurrence (local relapse or distant metastasis), DFS, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic evidence of ER/PR positive breast adenocarcinoma
2. Postmenopausal women.
3. Baseline LS and total hip BMD T-score > -2.0.
4. No prior treatment with denosumab or IV bisphosphonates is allowed.
5. No prior treatment with radiopharmaceuticals.
6. Not pregnant and not nursing.
7. Good dental health.
8. ECOG performance status 0-2.
9. Calculated creatinine clearance >= 30 mL/min.
10. Corrected serum calcium >= 8.0 mg/dL (2.00 mmol/L) and < 11.6 mg/dL (2.90 mmol/L)

Exclusion Criteria:

1. Patients with dental problems.
2. Patients with impaired renal functions
3. Patients with osteopenia, or T- score is below -2.0
4. Patients with history of serious drug hypersensitivity or drug allergy.

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenpausal women with ER/PR positive early breast cancer who are using adjuvant Letrozole
Enrollment: 50 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
The percentage change in lumber spine (L2-L4) BMD at 12 and 24 months for immediate- versus delayed-ZOL patients. | 24 months
  The percentage change in lumber spine (L2-L4) BMD at 12 and 24 months for immediate- versus delayed-ZOL patients.

SECONDARY OUTCOMES:
percentage change in total hip BMD at each assessment, fracture incidence in percentage, time to disease recurrence in months (local relapse or distant metastasis), DFS in months, and safety. | 24 months
  percentage change in total hip BMD at each assessment, fracture incidence in percentage, time to disease recurrence in months (local relapse or distant metastasis), DFS in months, and safety.
Fracture incidence in percentage | 24 months
  Assessment of incidence fracture in the participants

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Oncology Department, Assuit University Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 18 months